CLINICAL TRIAL: NCT02191904
Title: Laryngoscope Types and The Cervical Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Alkin Colak, Associate professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: alkin01
Record Dates: First submitted 2014-07-11; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Cervical Motion During Endotracheal Intubation

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Truview EVO2® (Active Comparator): Patients were randomly assigned into three groups with the sealed envelope method according to the laryngoscope type, which we had and we were used to; Macintosh type, Truview EVO2® type and Airtraq® type laryngoscopes were used in direct laryngoscopy Group DL (n=50), Truview EVO2® Group TV (n=50) and Airtraq® Group ATQ (n=50), respectively.
  Interventions: Other: Macintosh type, Truview EVO2® type and Airtraq® type laryngoscopes
- Airtraq® (Active Comparator): Patients were randomly assigned into three groups with the sealed envelope method according to the laryngoscope type, which we had and we were used to; Macintosh type, Truview EVO2® type and Airtraq® type laryngoscopes were used in direct laryngoscopy Group DL (n=50), Truview EVO2® Group TV (n=50) and Airtraq® Group ATQ (n=50), respectively
  Interventions: Other: Macintosh type, Truview EVO2® type and Airtraq® type laryngoscopes
- Direct laryngoscopy (Active Comparator): Patients were randomly assigned into three groups with the sealed envelope method according to the laryngoscope type, which we had and we were used to; Macintosh type, Truview EVO2® type and Airtraq® type laryngoscopes were used in direct laryngoscopy Group DL (n=50), Truview EVO2® Group TV (n=50) and Airtraq® Group ATQ (n=50), respectively
  Interventions: Other: Macintosh type, Truview EVO2® type and Airtraq® type laryngoscopes

INTERVENTIONS:
Other: Macintosh type, Truview EVO2® type and Airtraq® type laryngoscopes

SUMMARY:
To ensure minimal cervical motion during the intubation of trauma patients is important for the prevention of cervical spine injury (CSI) or further deterioration of existing CSI.

Intubation is required to secure the airway in patient during an anesthesia management or a mechanical ventilation at intensive care units. Laryngoscopes are the assisting tools for intubations. The most widely used laryngoscope type is one with a Macintosh blade. However, various types of laryngoscopes have been developed to be used for in case of difficult intubations, the intubation of the patients with head and neck trauma, or the intubation attempts carried out by inexperienced individuals. Truview EVO2® and Airtraq® are newly developed laryngoscopes, integrated with an optical view system.

The Truphatek TruView EVO2® (Truphatek International Ltd, Netanya, Israel) is a recently introduced, easy viewing type of laryngoscope, modified from the blades of Macintosh type laryngoscopes, having an angle of 46° at the end of blade and including a camera system that magnifies the image.

The Airtraq® laryngoscope (ATQ; King Medical Systems, Newark, DE) is also a newly developed type of laryngoscope, including optical imaging system. There is a channel on the device for the placement of the endotracheal tube. Endotracheal tube is inserted into the channel before the laryngoscopy. It has been reported that Airtraq is a novel single use laryngoscope which provides glottis display without any deviation in the normal position of the oral, pharyngeal or the tracheal axes.

In the literature, there are many studies comparing the effects of these newly developed laryngoscopes on cervical motions in different scenarios with cadavers and normal patients. However, in these studies, individual vertebral motion was reported during the placement of the tube, while the angulation of the head and neck and the difficulty of the intubations were not clear.

In this study our first hypothesis was cervical motion during endotracheal intubation in Truview EVO2® and Airtraq® types of laryngoscopes is lesser than Macintosh. The second one was the endotracheal intubation time is similar to the Macintosh that is used more often.

ELIGIBILITY:
Inclusion Criteria:

The patients who will undergo general anesthesia for abdominal surgery, American Society of Anesthesiologists physical status I to III, The patients who were aged between 20 and 75

Exclusion Criteria:

Our exclusion criteria were to have a history of emergency intubation or a difficult intubation, to have a body mass index higher than 35 or a rheumatologic disease that cause limitation of cervical motion, to have a previous history of cervical operation or tumor, trauma or infection on upper airway, and to have no tooth.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
CERVICAL MOTIONS | January 2011 and December 2012
  While the ventilation with face mask, different manupulations could be performed to the head. Therefore, neutral position was applied to the head before the laryngsocpy. In this procedure, the head was stabilized as the infraorbital edge and tragus is perpendicular to the ground. An inclinometer (A 360 degree angle gauge) was placed on the forehead of the patients, so that the tip of the inclinometer fits to glabellar line (figure 2,3). Inner diameter of the intubation tubes used for females and males were 7 to 7.5 mm and 8 to 8.5 mm, respectively. The maximum angulation were measured by an inclinometer and recorded from beginning of the laryngoscopy to the placement of the intubation tube into the trachea.

SECONDARY OUTCOMES:
Intubation Time | January 2011 and December 2012
  The duration between the beginning of the laryngoscope blade from passing the lips and the placement of the tube into trachea was recorded as intubation process time.

REFERENCES:
- [Derived] Colak A, Copuroglu E, Yilmaz A, Sahin SH, Turan N. A Comparison of the Effects of Different Types of Laryngoscope on the Cervical Motions: Randomized Clinical Trial. Balkan Med J. 2015 Apr;32(2):176-82. doi: 10.5152/balkanmedj.2015.15335. Epub 2015 Apr 1. PMID 26167342